CLINICAL TRIAL: NCT02402712
Title: Phase IIIb Study to Evaluate the Safety and Tolerability of Herceptin SC With Perjeta and Docetaxel in Patients With HER2-positive Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO29159; 2014-001458-40 (EudraCT Number)
Record Dates: First submitted 2015-03-23; First posted 2015-03-30 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; pertuzumab; Trastuzumab

ARMS (1):
- Herceptin SC + Perjeta IV + docetaxel IV (Experimental): Single arm
  Interventions: Drug: Docetaxel; Drug: pertuzumab [Perjeta]; Drug: trastuzumab [Herceptin]

INTERVENTIONS:
Drug: Docetaxel — Intravenous administration according to local label/clinical practice, after Herceptin and Perjeta.
Drug: pertuzumab [Perjeta] — Intravenous infusion every 3 weeks. First dose: 840 mg. Subsequent doses: 420 mg
  Other Names: RO4368451
Drug: trastuzumab [Herceptin] — Subcutaneous administration of 600 mg/5 mL every 3 weeks
  Other Names: RO0452317

SUMMARY:
This is an open-label, single-arm, multicenter, Phase IIIb study to evaluate the safety and tolerability of Herceptin SC in combination with Perjeta IV plus docetaxel in female patients with HER2-positive metastatic or locally recurrent breast cancer. Enrolled patients are to receive study medication until disease progression, unacceptable toxicity, withdrawal of consent, death, or predefined study end, whichever occurs first. The anticipated time on study treatment is approximately 24 months. The target sample size is 400.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed and documented adenocarcinoma of the breast with metastatic or locally recurrent disease not amenable to curative resection. Patients with measurable and/or non-measurable disease evaluable according to Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 are eligible.
* HER2-positive disease (defined as either immunohistochemistry [IHC] 3 + or in situ hybridization [ISH] positive) as assessed by local laboratory on primary tumor or metastatic site if primary tumor not available
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Left ventricular ejection fraction (LVEF) of at least 50%
* Negative serum pregnancy test result at baseline and use of effective contraception as defined by the protocol

Exclusion Criteria:

* Previous systemic non-hormonal anti-cancer therapy for the metastatic or locally recurrent disease. Note: Prior to study entry, up to two lines of hormonal therapy for metastatic or locally recurrent disease are permitted, one of which may be in combination with everolimus.
* Disease-free interval of less than 6 months from completion of adjuvant or neoadjuvant systemic non-hormonal treatment to recurrence of breast cancer
* Previous approved or investigative anti-HER2 agents as neoadjuvant or adjuvant therapy for any breast cancer treatment, except Herceptin
* History of persistent Grade 2 or higher hematological toxicity resulting from previous adjuvant or neoadjuvant therapy
* Radiographic evidence of central nervous system (CNS) metastases as assessed by computed tomography (CT) or magnetic resonance imaging (MRI), unless they have been treated and have been stable for at least 3 months and do not require ongoing corticosteroid treatment
* Current peripheral neuropathy of Grade 3 or greater
* History of other malignancy within the last 5 years prior to first dose of study drug administration, except for carcinoma in situ of the cervix or basal cell carcinoma
* Inadequate organ function
* Uncontrolled hypertension with or without medication
* Clinically significant cardiovascular disease
* History of LVEF decline to below 50% during or after prior Herceptin neo-adjuvant or adjuvant therapy
* Current known infection with HIV, hepatitis B virus, or hepatitis C virus
* Severe uncontrolled concomitant disease that would contraindicate the use of any of the investigational drugs used in this study or that would put the patient at high risk for treatment-related complications, including severe pulmonary conditions/illness
* Pregnant or lactating women
* Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy
* History of receiving any investigational treatment within 28 days prior to first dose of study drug administration (dosing) or concurrent participation in any interventional clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 24 months after the last patient has been enrolled, approximately 3.5 years
Incidence and severity of adverse events Grade >/= 3, according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.0 | Up to 24 months after the last patient has been enrolled, approximately 3.5 years
Incidence of cardiac events (composite outcome measure): congestive heart failure (CHF) and cardiac death | Up to 24 months after the last patient has been enrolled, approximately 3.5 years

SECONDARY OUTCOMES:
Progression-free survival, tumor assessments according to RECIST v1.1 | Up to 3.5 years
Overall survival | Up to 3.5 years
Objective response rate, defined as a complete response (CR) or a partial response (PR) | Up to 3.5 years
Incidence of anti-Herceptin, anti-rHuPH20 antibodies | Up to 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (112):
- Belgium (6):
  - AZ Sint Jan, Bruges
  - UZ Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - CHU Sart-Tilman, Liège
  - Clinique Saint-Joseph, Liège
  - Sint Augustinus Wilrijk, Wilrijk
- Bulgaria (7):
  - Multiprofile Hospital For Active Treatment Dr. Tota Venkova JSC, Gabrovo
  - Multiprofile Hospital for Active Treatment Central Onco Hospital OOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Comprehensive Cancer Center-Plovdiv, Plovdiv
  - Specialized Hospital for Active Treatment of Oncological Diseases - Sofia District EOOD, Sofia
  - Specialized Hospital for Active Cancer Treatment, Dr. Mark Antonov Markov - Varna Ltd, Varna
  - MDOZS Vrasta Ltd., Vratsa
- Canada (2):
  - Moncton Hospital, Moncton, New Brunswick
  - Royal Victoria Regional Health Centre, Barrie, Ontario
- France (14):
  - Centre Hospitalier Regional Metz-Thionville - Hopital de Mercy, Ars-Laquenexy
  - Medipole De Savoie; Departement Oncologie, Challes-les-Eaux
  - Hopital Prive Sainte Marie, Chalon-sur-Saône
  - Centre Hospitalier Louis Pasteur, Chartes Le Coudray
  - Pole Sante Republique; Pharmacie Oncologique, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - CHU de Grenoble, Grenoble
  - Hopital Europeen, Marseille
  - Centre Hospitalier de Mont de Marsan - Hopital Layne, Mont-de-Marsan
  - Hopital Saint Joseph; Service de Rhumatologie, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Strasbourg Oncologie Libérale, Strasbourg
  - Gustave Roussy, Villejuif
- Germany (14):
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - Onkologische Schwerpunktpraxis Dr. Joerg Schilling, Berlin
  - Universitaetsklinikum Erlangen, Erlangen
  - Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Essen, Essen
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Universitatsklinikum Schleswig-Holstein; Klinik fuer Innere Medizin I, Lübeck
  - Onkologische Schwerpunktpraxis Lübeck, Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Suedharz Klinikum Nordhausen gGmbH, Nordhausen
  - Sana Klinikum Offenbach GmbH; Klinik für Gynäkologie & Geburtshilfe, Offenbach
  - Johanniter-Krankenhaus Genthin - Stendal GmbH; Gynäkologie und gynäkologische Onkologie, Stendal
  - Klinikum Mutterhaus der Borromaeerinnen, Trier
  - Universitätsklinikum Würzburg, Würzburg
- Hungary (7):
  - Szent Margit Hospital; Dept. of Oncology, Budapest
  - Ogyi, Orszagos Gyogyszereszeti Intezet, Budapest
  - Semmelweis Egyetem, Budapest
  - Szent Imre Egyetemi Oktatokorhaz, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont; Fázis I-es Klinikai Farmakológiai Vizsgálóhely, Budapest
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház, Miskolc
- Italy (21):
  - Azienda Ospedaliera Regionale San Carlo, Potenza, Basilicate
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori, Meldola, Emilia-Romagna
  - Azienda Ospedaliero - Universitaria di Modena Policlinico, Modena, Emilia-Romagna
  - Azienda Ospedaliera di Reggio Emilia - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Ospedale Infermi di Rimini, Rimini, Emilia-Romagna
  - Istituti Fisioterapici Ospitalieri, Rome, Lazio
  - Ospedale Policlinico San Martino, Genoa, Liguria
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - Asst Della Valtellina E Dell'Alto Lario, Sondrio, Lombardy
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele, Catania, Sicily
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli, Tuscany
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda USL 5 di Pisa, Pisa, Tuscany
  - Ospedale Santo Stefano, Azienda USL Centro Prato, Prato, Tuscany
  - Azienda Ospedaliera Santa Maria di Terni, Terni, Umbria
  - Azienda Ospedaliero-Universitaria di Ferrara, Arcispedale Sant'Anna, Cona (Ferrara), Veneto
  - Ospedale Sacro Cuore Don Calabria, Negrar, Veneto
  - IOV - Istituto Oncologico Veneto IRCCS, Padua, Veneto
  - "Azienda Ospedaliera Universitaria Integrata Verona Ospedale Borgo Trento", Verona, Veneto
- Mexico (6):
  - Consultorio de Medicina Especializada, México, Mexico CITY (federal District)
  - Grupo Medico Camino, DF
  - Superare Centro de Infusion S.A. de C.V., México
  - Fundacion de Cancer de Mama.A.C., México
  - Centro Medico San Jose, Monterrey, Nuevo Leon
  - Cancerología, Querétaro
- Poland (13):
  - Bialostockie Centrum Onkologii im. Marii Sklodowskiej - Curie, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Copernicus Podmiot Medyczny Sp. z o.o. Wojewodzkie Centrum Onkologii, Gdansk
  - Szpitale Pomorskie Sp. z o. o., Gdynia
  - Przychodnia Lekarska KOMED, Konin
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Onkologii Ziemi Lubelskiej im. św. Jana z Dukli, Lublin
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej MSW z W-MCO w Olsztynie, Olsztyn
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Opolskie Centrum Onkologii, Opole
  - Szpital Kliniczny; Przemienienia Panskiego;Uniwersytetu Medyczny im.; Karola Marcinkowskiego w Pozna, Poznan
  - Wielkopolskie Centrum Onkologii, Poznan
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie; Klinika Onkologiczna, Warsaw
  - MAGODENT Sp. z o.o., Warsaw
- Portugal (5):
  - Hospital de Braga, Braga
  - Instituto Portugues Oncologia de Coimbra Francisco Gentil, EPE, Coimbra
  - Hospital da Luz, Lisbon
  - Centro Hospitalar de Lisboa Norte, EPE - Hospital Santa Maria, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Spain (7):
  - Complexo Hospitalario Universitario de Santiago (CHUS) - Hospital Clinico Universitario, Santiago de Compostela, LA Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Fundacion Instituto Valenciano de Oncologia (IVO), Valencia
- United Kingdom (10):
  - Betsi Cadwaladr University Health Board, Bangor Gwynedd
  - Velindre Cancer Centre, Cardiff
  - Dorset County Hospital, Dorchester
  - University Hospitals of Leicester NHS Trust - Leicester Royal Infirmary, Leicester
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Mount Vernon Cancer Centre, Northwood
  - Peterborough City Hospital, Peterborough
  - Portsmouth Hospitals NHS Trust - Queen Alexandra Hospital, Portsmouth
  - Royal Cornwall Hospitals NHS Trust, Truro

REFERENCES:
- [Derived] Kuemmel S, Tondini CA, Abraham J, Nowecki Z, Itrych B, Hitre E, Karaszewska B, Juarez-Ramiro A, Morales-Vasquez F, Perez-Garcia JM, Cardona-Huerta S, Monturus E, Sequi M, Restuccia E, Benyunes M, Martin M. Subcutaneous trastuzumab with pertuzumab and docetaxel in HER2-positive metastatic breast cancer: Final analysis of MetaPHER, a phase IIIb single-arm safety study. Breast Cancer Res Treat. 2021 Jun;187(2):467-476. doi: 10.1007/s10549-021-06145-3. Epub 2021 Mar 21. PMID 33748921